CLINICAL TRIAL: NCT01511367
Title: A Double-blind, Double Dummy, Randomised, Parallel Group, Multicentre Study to Compare the Efficacy and Safety of Flutiform pMDI With Fluticasone pMDI and With Seretide pMDI in Paediatric Subjects Aged 5 to Less Than 12 Years With Moderate to Severe Persistent Reversible Asthma
Brief Title: Comparison of Flutiform, Fluticasone and Seretide in Treatment of Moderate to Severe Asthma in Paediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FLT3506; 2010-024635-16 (EudraCT Number)
Record Dates: First submitted 2011-12-07; First posted 2012-01-18 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Asthma
Keywords: moderate to severe persistent reversible asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone-formoterol; Fluticasone-Salmeterol Drug Combination; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Flutiform (Active Comparator)
  Interventions: Drug: Flutiform
- Seretide (Active Comparator)
  Interventions: Drug: Seretide
- Flixotide (Active Comparator)
  Interventions: Drug: Flixotide

INTERVENTIONS:
Drug: Flutiform — 50/5ug (fluticasone/formoterol) 2 puffs twice daily
  Arms: Flutiform
Drug: Seretide — 50/25 ug (fluticasone/salmeterol) 2 puffs twice daily
  Arms: Seretide
Drug: Flixotide — 50ug 2 puffs twice daily
  Arms: Flixotide

SUMMARY:
This is a comparator study to assess safety and efficacy of Flutiform compared with Fluticasone pMDI and Seretide pMDI in paediatric asthma patients with moderate to severe persistent, reversible asthma.

DETAILED DESCRIPTION:
This is a study involving a 2-4 week run-in phase followed by a 12 week double blind treatment phase. During the run-in phase, all subjects receive Flixotide. In the treatment phase subjects will be randomised to one of the 3 treatment groups and will receive active Flutiform and placebo Flixotide or Active Seretide and placebo Flixotide or active Flixotide and either placebo seretide or placebo Flutiform. Efficacy will be assessed by lung function tests, asthma symptoms, sleep disturbance due to asthma and rescue medication use. Safety will be assessed by adverse events, lab tests, urinary cortisol and vital signs.

ELIGIBILITY:
Inclusion Criteria

1. Male and Female subjects 5 to <12 years old.
2. Known history of moderate to severe persistent reversible asthma1 for ≥ 6 months prior to the screening visit.
3. Demonstrated FEV1 of ≥ 60% to ≤ 90% for predicted normal values (Polgar 1971) during the screening period following appropriate withholding of asthma medications (if applicable):

   * No LABA use within 12 hours and/or no SABA use within 6 hours of the PFT
   * No use of inhaled ICS-LABA asthma therapy within 12 hours of the PFT
   * Inhaled corticosteroids are allowed on the day of screening
4. Documented reversibility of ≥ 15% in FEV1 in the screening period
5. Current use of an inhaled corticosteroid for asthma at a stable dose for at least 4 weeks prior to the screening visit
6. Inadequate asthma control on an ICS alone at a dose of ≤ 500 µg fluticasone equivalents/day, OR controlled asthma on an ICS-LABA combination at a ICS dose of ≤ 200 µg fluticasone equivalents/day
7. Demonstrated satisfactory technique in the use of the pMDI and spacer device
8. Can perform spirometry adequately
9. Willing and able to enter information in the electronic diary with the help of a parent or guardian, if necessary and attend all study visits
10. Willing and able to substitute pre-study prescribed inhaled asthma medication for the entire duration of the study
11. If a female subject is post menarche a urine pregnancy test may be undertaken at the discretion of the investigator and the subjects' parent(s) /legal representative. This test must be negative.
12. Written informed consent and assent obtained as per national law

Exclusion Criteria

1. Near fatal or life-threatening (including intubation) asthma within the past year
2. Hospitalisation or an emergency visit for asthma within the past 6 months
3. History of systemic (injectable or oral) corticosteroid medication within 1 month of the screening visit
4. Current or prior non-response or partial response only to an ICS-LABA combination1
5. Evidence of a clinically unstable disease, as determined by medical history, clinical laboratory tests, and physical examination that, in the Investigator's opinion, preclude entry into the study. "Clinically significant" is defined as any disease that, in the opinion of the Investigator, would put the subject at risk through study participation, or which would affect the outcome of the study
6. In the Investigator's opinion a clinically significant upper or lower respiratory infection within 4 weeks prior to the screening visit
7. Significant, non-reversible active pulmonary disease (e.g. cystic fibrosis, bronchiecstasis, tuberculosis)
8. Known Human Immunodeficiency Virus (HIV)-positive status
9. Current smoking history within 12 months prior to the screening visit
10. Current evidence of alcohol or substance abuse within 12 months prior to the screening visit
11. Subjects who have taken β- blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrythmics, or potent CYP 3A4 inhibitors such as ketoconazole within 1 week prior to the screening visit
12. Current use of medications, other than those allowed in the protocol, that in the investigator's opinion will have an effect on bronchospasm and/or pulmonary function
13. Current evidence of hypersensitivity or idiosyncratic reaction to test medications or components
14. Receipt of an Investigational medicinal product within 30 days of the screening visit
15. Current participation in a clinical study

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 498 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To show superiority in the efficacy of Flutiform pMDI 50/5μg (2 puffs bid) versus fluticasone pMDI 50 μg (2 puffs bid). | 12 weeks
  Change from pre-dose Forced Expiratory Volume in one second (FEV1) in litres at baseline to 2 hours post-dose FEV1 at the end of the 12 week treatment period.

SECONDARY OUTCOMES:
Show non-inferiority in the efficacy of Flutiform to Seretide | 12 weeks
  Change from pre-dose FEV1 at baseline to 2 hours post-dose FEV1 at Day 1 and FEV1 AUC0-4 at Day 1 and Week 12 (Flutiform vs Seretide)

CONTACTS AND LOCATIONS:
Locations (8):
- Plovdiv, Bulgaria
- Alergologie Skopkova s.r.o, Ostrava-Marianske Hory, Czechia
- Illés és Ádám Egészségügyi Szolgáltató Bt., Kiskunhalas, Hungary
- New Dehli, India
- Alergo-Med Specjalistyczna Przychodnia Lekarska Sp.z.o.o., Tarnów, Poland
- Spitalul Judetean de Urgenta Deva, Deva, Hunedoara, Romania
- Moscow, Russia
- Odesa, Ukraine

REFERENCES:
- See also: Link to Results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT3506